CLINICAL TRIAL: NCT05571878
Title: Is Brain Insulin Resistance a Feature of the Biology of Depression: a Pilot Multi-modality Neuroimaging Study in Adolescents
Brief Title: Is Brain Insulin Resistance a Feature of the Biology of Depression in Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 030/2020
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder; Depression
Keywords: Major Depressive Disorder; Insulin Resistance; Type 2 Diabetes; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Intervention Model Description: The study will follow a single blind, crossover design wherein each participant will complete an MRI based protocol of brain insulin action. After an overnight fast, fasting bloodwork will be obtained, followed by two MRI scans: one with intranasal placebo and one with intranasal insulin challenge (80 IU; 40 IU per nostril). Between scans they will have a short break and be asked to complete a cognitive assessment. Participants with depression will complete a 6-month follow-up visit to track changes in metabolic health, illness severity, and cognitive function.
Masking Description: Participants will be blinded to the order of the intranasal spray condition (insulin or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Crossover: Insulin and Placebo (Experimental): Twelve adolescents who have a confirmed depression diagnosis or experiencing depression will be used as the study population group against 12 healthy adolescents who will be used as the healthy study population group.
  Both the health control group and medication-free adolescents with depression will receive the same drug conditions (intranasal insulin and intranasal placebo).
  Interventions: Drug: Humalog; Drug: Saline nasal spray

INTERVENTIONS:
Drug: Humalog — All participants will be given an intranasal insulin challenge (80 IU) to assess brain insulin signalling via MRI based assay
  Other Names: Intranasal Insulin
Drug: Saline nasal spray — All participants will be given an intranasal saline placebo (0.8 mL) in order to establish baseline brain insulin signalling via MRI based assay
  Other Names: Intranasal Placebo

SUMMARY:
This study will examine if brain insulin resistance is a feature of depression in humans using magnetic resonance imaging (MRI) measures sensitive to brain insulin action. This study will examine adolescents, as depression onset commonly occurs during this age, and the impacts of cumulative medication exposure and other lifestyle-related confounds are also lower in this age group, improving our ability to understand the underlying biology.

DETAILED DESCRIPTION:
BACKGROUND: Major depressive disorder (MDD) is associated with metabolic dysfunction, including higher body mass index and increased risk for type 2 diabetes (T2D). This relationship is bidirectional as insulin resistance is associated with greater depressive symptom severity and worse cognition. These nested relationships between metabolic and mental health have encouraged a reconceptualization of MDD as a metabolic disorder. In this context, insulin in the brain has been implicated as a potential mediator unifying the mechanisms underlying metabolic and mental health. There is early evidence supporting this hypothesis; mice with brain-specific knockout of insulin receptor exhibited depression-like behavior that was reversed by treatment with monoamine oxidase inhibitors, while anti-diabetic agents that can potentially cross the blood-brain barrier have shown initial promise in reducing depressive symptoms.

HYPOTHESES: 1) Adolescents diagnosed with MDD will have greater brain insulin resistance in comparison to matched healthy controls. 2) Greater brain insulin resistance will be associated with increased illness severity, worse cognitive performance, and worse short-term outcomes (i.e., at 6 months) in the depression group. 3) Greater peripheral insulin resistance (measured using fasting blood work) and hepatic and visceral adiposity (measured using MRI) will be associated with greater brain insulin resistance.

APPROACH AND METHODOLOGY: Twelve adolescents with depression (14 to 18 years old) and 12 age-, sex-, and BMI-matched healthy controls will be recruited for the study. In a single-blinded crossover design, all 24 participants will undergo fasting blood work (glucose, insulin, and c-peptide) followed by an MRI-based protocol of brain insulin action. This includes two MRI scans; one with intranasal insulin challenge (80 IU) and one with intranasal placebo. This protocol leverages the property of intranasal insulin to induce resting state connectivity and blood flow changes in the brain. This will be achieved using a 3 Tesla (3T) MRI scanner, where participants will undergo a high-resolution T1-weighted structural scan, a resting state functional MRI scan, and an arterial spin labeling scan. Single voxel 1H-magnetic resonance spectroscopy will also be employed to examine changes in glutamate levels in the frontal and temporal cortex. The difference in change induced by intranasal insulin compared to that with intranasal placebo will be utilized as an index of insulin activity since any difference observed between placebo and insulin during this controlled manipulation is likely to be due to the intranasal insulin. THINC-it, a brief cognitive assessment, will also be performed to measure cognitive function in relation to insulin induced brain changes. An abdominal surface coil scan will also be used to measure visceral and hepatic adiposity. Participants with depression will be invited for a six-month follow-up visit to repeat fasting blood work, along with clinical and cognitive assessments. Age, sex, and BMI will be used as covariates in all analyses.

SIGNIFICANCE: Demonstrating disrupted brain insulin action can provide novel insights into poorly understood mechanisms underlying the relationship between MDD and T2D. Evidence of brain insulin resistance early in the course of illness may also identify a modifiable risk factor that can be targeted using brain insulin sensitizers at the earliest stages of the illness. Thus, this work that lies at the intersection of psychiatry, physiology, and psychopharmacology has the potential to generate new knowledge and improve outcomes in an area of significant unmet need.

ELIGIBILITY:
Inclusion Criteria:

* Age 14- 18
* One of the following: Diagnosis of Major Depressive Disorder (MDD) or Persistent Depressive Disorder (PDD); or score ≥22 on the Mood and Feeling Questionnaire and confirmation of depression with the Mini International Neuropsychiatric Interview Kid (MINI Kid)
* BMI between 5-95th population percentile and Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) ≤2.5 calculated using fasting blood work values (glucose and insulin)

Exclusion Criteria:

* History of primary psychotic illness
* Use of antipsychotics or mood stabilizers
* History of current substance use disorder (moderate to severe)
* Pre-diabetes or diabetes (fasting glucose ≥6.0 mmol/l or use of anti-diabetic drug)
* Evidence of impaired glucose tolerance on screening oral glucose tolerance test (OGTT)
* Use of weight, lipids, or blood pressure reducing agents
* History of liver disease or AST>2 times upper limit of normal
* History of kidney disease
* MRI contraindications
* Positive pregnancy test
* Allergic to exogenous insulin
* Positive result on urine drug screen (participants with positive cannabis and alcohol urine drug screens may still be eligible for the study; positive drug screens for other substances will be exclusionary)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
The change in brain imaging outcomes, measuring brain insulin resistance, following intranasal insulin or placebo challenges, compared between the participants with depression and healthy controls. | Study Visit 1- MRI #1 15 minutes after intranasal challenge #1, MRI #2 15 minutes after intranasal challenge #2
  Brain insulin resistance will be measured by changes in fMRI, 1H- MRS, and ASL measured during MRI scans following intranasal insulin and placebo challenge. These changes will be compared within subjects and between groups (depression vs controls).
  1. Resting state functional MRI (fMRI) will measure connectivity between prefrontal brain regions and hippocampus.
  2. Single voxel proton magnetic resonance spectroscopy (1H- MRS) will measure the glutamate levels in the temporal and frontal cortex.
  3. Arterial spin labeling (ASL) will be used to measure cerebral blood flow in the hypothalamus and the prefrontal cortex.

SECONDARY OUTCOMES:
Correlation between brain insulin resistance with illness severity and cognitive functioning at baseline and 6-month study follow up | Illness Severity: Study Visit 1, pre-intervention (MRI scan #1), and 6-month follow-up study visit following fasting blood work; Brain Insulin Resistance: Study Visit 1, during MRI scan #1 and #2
  Primary outcome measures will be used to assess the correlation between brain insulin resistance (MRI measures; described in Outcome 1) and illness severity.
  Illness Severity- Center for Epidemiological Studies- Depression Scale for Children (CES-DC). 20 item self-report depression inventory with possible scores ranging from 0-60. Higher scores are indicative of worse illness severity. A cut-off score of 15 is suggestive of depressive symptoms in children and adolescents.
Correlation between brain insulin resistance with cognitive functioning at baseline and 6-month study follow up | Cognitive Function: Study Visit 1, during break between MRI scan #1 and #2, and 6-month follow-up study visit following fasting blood work; Brain Insulin Resistance: Study Visit 1, during MRI scan #1 and #2
  Primary outcome measures will be used to assess the correlation between brain insulin resistance (MRI measures; described in Outcome 1) with cognitive functioning.
  Cognitive Functioning- THINC-it® (interactive cognitive assessment tool). Brief screening tool designed to measure cognition and determine whether cognitive functioning is impaired. Higher score is indicative of better performance, scores can range from 0-4000.

OTHER OUTCOMES:
Correlation between brain insulin resistance and peripheral insulin resistance at baseline and 6-month study follow up | Peripheral Insulin Resistance: Study Visit 1, pre-MRI #1 and post-MRI #2, and 6-month follow-up study visit; Brain Insulin Resistance: Study Visit 1, during MRI scan #1 and #2
  Primary outcome measures will be used to assess the correlation between brain insulin resistance (MRI measures; described in Outcome 1) with peripheral insulin resistance.
  Peripheral Insulin Resistance - Fasting bloodwork: Glucose (mmol/L), insulin (pmol/L), C-peptide (pmol/L).
Correlation between brain insulin resistance, and hepatic and visceral adiposity | Hepatic and Visceral Adiposity: Study Visit 1, during MRI #1; Brain Insulin Resistance: Study Visit 1, during MRI scan #1 and #2
  Primary outcome measures will be used to assess the correlation between brain insulin resistance (MRI measures; desired in Outcome 1) with hepatic and visceral adiposity
  Hepatic and Visceral Adiposity- Abdominal MRI Scan (cm^3)

CONTACTS AND LOCATIONS:
Overall Officials: Mahavir Agarwal, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No